CLINICAL TRIAL: NCT01522404
Title: A 6 Month, Phase II Randomized, Double-Blind, Placebo Controlled, Flexible Dosing, Crossover Trial of Atomoxetine in Subjects With Mild Cognitive Impairment.
Brief Title: Effects of Atomoxetine in Mild Cognitive Impairment
Acronym: ATX-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Allan I Levey, MD, Professor and Chair, Department of Neurology, Emory University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00054397; 5U01AG010483 (NIH); ATX-001 (Other: Other)
Record Dates: First submitted 2012-01-25; First posted 2012-01-31 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Memory Loss; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Alzheimer Disease | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atomoxetine / Inactive Compound (Experimental): Participants in this arm received atomoxetine, starting with 10 mg po daily and increasing weekly by increments to a maximum of 100 mg po daily or the maximum tolerated dose for up to weeks 29 and are then crossed over to Inactive compound group
  Interventions: Drug: Atomoxetine; Drug: Placebo
- Inactive compound / Atomoxetine (Placebo Comparator): Subjects in this arm received a matching placebo that have inactive compound for up to weeks 29 and then are crossed over to receive active treatment of Atomoxetine
  Interventions: Drug: Atomoxetine; Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Subjects in this intervention will receive Atomoxetine up to 29 weeks, crossover, dose escalating (up to a maximum dose of 100 mg per day) of oral atomoxetine
  Other Names: Strattera; Primary Outcome Measure
Drug: Placebo — Subjects in this intervention will receive inactive compound up to weeks 29 and will cross over to the other group
  Other Names: Inactive compound

SUMMARY:
The purpose of this study is to evaluate the safety of atomoxetine and its effect primarily on the biologic markers (substances that may indicate the presence of a disease) in the cerebrospinal fluid (CSF) of participants diagnosed with Mild Cognitive Impairment (MCI). Additionally, information will be gathered to identify the dose of atomoxetine that is most beneficial, and how taking this medication affects thinking and behavior, as well as imaging and blood biomarkers.The study will also explore rates of change in biomarkers of neurodegeneration (Aß, tau, brain atrophy rates). The results of this research will help determine if atomoxetine alters signs of inflammation and other biomarkers associated with Alzheimer's disease.

DETAILED DESCRIPTION:
The Alzheimer's Disease (AD) epidemic is a looming crisis, with an urgent need for new therapies to delay or prevent symptom onset and progression. Advances in AD biomarker research have demonstrated changes in amyloid, brain metabolism, and other pathophysiologies prior to the onset of memory loss, with some markers possibly changing one or two decades earlier. Since MCI coincides with the onset of brain atrophy, this early stage of AD pathogenesis may offer a critical window of time to initiate novel therapies aimed at the secondary wave of events that lead to progressive neurodegeneration.

From recently emerged basic research in animal models of AD: loss of norepinephrine (NE) incites a pro-inflammatory condition that is neurotoxic and reduces Aß clearance, and remarkably, rescue of norepinephrine reverses these effects and slows neurodegeneration. This study seeks to extend this proof-of-concept to humans for the first time. The study proposes that atomoxetine, a selective norepinephrine transport inhibitor, is an ideal drug to translate these findings to humans because it is already FDA-approved and safe in the elderly

Subjects with mild cognitive impairment (amnestic or multi-domain subtypes) will be randomly assigned to treatment with placebo or flexible doses of the Norepinephrine Transporter (NET) inhibitor atomoxetine, starting with 10 mg po daily and increasing weekly by increments to a maximum of 100 mg po daily or the maximum tolerated dose. Participants will be treated for upto 29 weeks, and will undergo venous blood draws and lumbar puncture for biomarker analyses at baseline and up to weeks 29. At a maximum of 29 weeks time point, subjects assigned to active treatment will crossover to placebo and those subjects who were initially randomized to placebo will initiate active treatment.

Participants who complete study are eligible to receive open-label Atomoxetine at the maximum-tolerated dose received during the double-blind phase of the trial. Subjects in the open label are seen every at week 29 upto maximum of 2 years.

ELIGIBILITY:
Inclusion

* Subjects must have a subjective memory concern as reported by subject, study partner or clinician.
* Meets Alzheimer's Disease Neuroimaging Initiative (ADNI) criteria for diagnosis of MCI. Subjects with amnestic (single or multi-domain) will be eligible, as both subtypes of MCI are at high risk for progression to AD.
* Abnormal memory function documented by assessment using the Logical Memory subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale-Revised (the maximum score is 25):

  * <11 for 16 or more years of education
  * <9 for 8-15 years of education
  * <6 for <7 years of education
* Mini-Mental State Exam score between 24 and 30 (inclusive). Exceptions may be made for subjects with less than 8 years of education at the discretion of the PI.
* Clinical Dementia Rating = 0.5. Memory Box score must be at least 0.5.
* General cognition and functional performance sufficiently preserved such that a diagnosis of AD cannot be made by the physician at the time of the screening visit.
* Cholinesterase inhibitors and memantine are allowable if stable for 12 weeks prior to screen.
* Stability of Permitted Medications for 4 weeks. In particular, subjects may washout from excluded medication for at least 4 weeks prior to screening.
* Geriatric Depression Scale (GDS) ≤ than 6.
* Male or female outpatients aged 50-90 (inclusive).
* Study partner has regular contact with the subject adequate to provide a reliable assessment of the subject's level of function, and can be available for all clinic visits, either in person or by telephone, for the duration of the study.
* Visual and auditory acuity adequate for neuropsychological testing.
* Good general health with no diseases expected to interfere with the study.
* For women of child-bearing potential (i.e., one who is biologically capable of becoming pregnant), must be willing to use a medically acceptable form or birth control or practice abstinence for the duration of her participation in the trial. Acceptable methods of birth control include: oral or patch contraception, or medroxyprogesterone (Depo-Provera®) or other intramuscular contraceptive injection, or implantation of levonorgestrel (Norplant®) system, an Intrauterine Device (IUD), a reliably-employed barrier method (e.g. diaphragm, cervical cap or condom), or a male partner who is surgically sterilized.
* Modified Rosen Hachinski ≤ 4.
* Completed six grades of education or has a good work history (sufficient to exclude mental retardation).
* Able to communicate in English with study personnel.
* Able to understand the nature of the study and must provide written informed consent prior to conduct of any study procedures.
* Willing to undergo repeated MRIs (3Tesla) and at least three Positron-Emission Tomography (PET) scans. No medical contraindications to MRI.
* Agrees to blood collection for Apolipoprotein (APOE) epsilon, CYP2D6 and biomarker testing.
* Agrees to lumbar puncture over the course of the study for the collection of CSF. CSF levels of Ab42, total Tau, and Tau phosphorylated at threonine 181 consistent with underlying AD pathology according to established threshold values at Emory and the ADNI Biomarker Core

Exclusion

* Any significant neurologic disease other than MCI and suspected incipient AD, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, poorly controlled seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
* Screening/baseline MRI scan with evidence of infection, large vessel infarction or other focal structural lesions that could account for the memory deficits. Subjects with multiple lacunes or lacunes in a critical memory structure are excluded.
* Contraindication to MRI due to presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, or excessive weight.
* Presence of clinically significant suicide risk, based on the Investigator's judgment informed by a structured clinician interview. Any suicide attempt within the past 1 year of the screening visit is exclusionary.
* Major depression, bipolar disorder as described in DSM-IV within the past 1 year, or history of schizophrenia (DSM-IV). Psychotic features, agitation or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol.
* History of alcohol or substance abuse or dependence within the past 2 years (DSM-IV criteria).
* Allergic to any component of atomoxetine (Strattera).
* Any uncontrolled medical condition that is expected to preclude completion of the study, or any medical condition which would represent a contraindication to atomoxetine pharmacotherapy (e.g. hepatic insufficiency, untreated hypertension, untreated cardiovascular or cerebrovascular disease).
* Known serious structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, or other serious cardiac problems.
* History of narrow angle glaucoma.
* History of pheochromocytoma.
* Clinically significant abnormal findings on screening laboratory tests or physical exam. Abnormalities in Vitamin B12 level, Thyroid Function Tests (TFTs) or Liver Function Tests (LFTs) that might interfere with the study. A low Vitamin B12 level is exclusionary, unless follow-up labs (homocysteine and methylmalonic acid indicate that it is not physiologically significant.
* Slow metabolizer of atomoxetine (i.e., CYP2D6 polymorphism).
* Women who are pregnant or lactating, or who plan to become pregnant during the study.
* Current use of warfarin (exclusionary for lumbar puncture).
* Inability to obtain initial CSF sample.
* Use within 60 days of a monoamine oxidase inhibitor or a potent CYP2D6 inhibitor.
* Current use of anti-psychotic medication.
* Current use of the following anti-depressant medications that act on NET: duloxetine, venlafaxine, desvenlafaxine, imipramine, or amitryptiline.
* Current participation in another clinical trial. Participation in clinical studies involving neuropsychological measures being collected more than one time per year.
* CSF profile is not consistent with underlying Alzheimer's Disease pathology.
* Reasonable likelihood for non-compliance with the protocol or any other reason, in the opinion of the investigator, prohibits enrollment of subject into the study.
* Exceptions to these guidelines may be considered on a case-by-case basis at the discretion of the protocol director.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan I. Levey, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between March 2012 and October 2017. The study is conducted at Emory University Hospital in Atlanta.
Groups:
- Atomoxetine / Inactive Compound: Participants in this group are randomized to Atomoxetine, starting with 10 mg po daily and increasing weekly by increments to a maximum of 100 mg po daily or the maximum tolerated dose during period 1/ Matching placebo that have inactive compound during period 2.
- Inactive Compound / Atomoxetine: Participants in this group are randomized to matching placebo that have inactive compound during period 1/ Atomoxetine, starting with 10 mg po daily and increasing weekly by increments to a maximum of 100 mg po daily or the maximum tolerated dose during period 2.
Period: First Intervention (up to Week 29)
Arm/Group | Atomoxetine / Inactive Compound | Inactive Compound / Atomoxetine
Started | 20 | 19
Completed | 18 | 19
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Second Intervention (up to Week 58)
Arm/Group | Atomoxetine / Inactive Compound | Inactive Compound / Atomoxetine
Started | 18 | 19
Completed | 17 | 19
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine / Inactive Compound | Inactive Compound / Atomoxetine | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (5.7) | 72.0 (7.5) | 71.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Interleukin 1 (IL 1-alpha) in Cerebrospinal Fluid (CSF) in Subjects With Mild Cognitive Impairment (MCI) Treated With Atomoxetine/Inactive Compound Compared to Subjects Treated With Inactive Compound / Atomoxetine
Description: This study will examine the effects of Atomoxetine and Inactive compound on biomarkers of inflammation by measuring and comparing the levels of Interleukin 1 (IL 1-alpha) using the assay of CSF at Baseline, Week 29 and Week 58 among the two groups. The study hypothesizes that the period that participants are treated with atomoxetine will have reductions in levels of these pro-inflammatory biomarkers among the two groups.
Time Frame: Baseline, Week 29 and Week 58
Population: Only 15.1 % of the samples were above the limit of detection for Interleukin 1 (IL 1-alpha) alpha in CSF, precluding the planned analysis and comparing the mean and standard deviation of Interleukin 1 (IL 1-alpha) alpha levels in treatment versus placebo groups. Hence the analysis was not done and the outcome was not measured.
Arm/Group | Atomoxetine / Inactive Compound | Inactive Compound / Atomoxetine
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Mean Level of Thymus-Expressed Chemokine (TECK) in Cerebrospinal Fluid (CSF) in Participants With Mild Cognitive Impairment (MCI) Treated With Atomoxetine / Inactive Compound Compared to Participants Treated With Inactive Compound / Atomoxetine
Description: This study will examine the effect of Atomoxetine and Inactive Compound on biomarkers of inflammation by measuring and comparing the mean levels of Thymus-Expressed Chemokine (TECK). These levels are measured using the assay of CSF at Baseline, Week 29 and Week 58. The study hypothesizes that the period that participants are treated with atomoxetine will have reduction in levels of these markers among both groups.
Time Frame: Baseline, Week 29 and Week 58
Population: Only 49.1 % of the samples were above the limit of detection for TECK in CSF among the groups that are included in the analysis below. The levels for only 18 participants in Atomoxetine group and 18 participants in Inactive compound were analyzed
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Atomoxetine: Participants in this group received Atomoxetine, starting with 10 mg po daily and increasing weekly by increments to a maximum of 100 mg po daily or the maximum tolerated dose.
- Inactive Compound / Placebo: Participants in this group receive matching placebo that have inactive compound
Arm/Group | Atomoxetine | Inactive Compound / Placebo
Number analyzed (Participants) | 18 | 18
pg/mL
  Baseline | 1 (0.4) | 0.8 (0.2)
  Week 29 | 1 (0.4) | 0.9 (0.2)
  Week 58 | 1.1 (0.7) | 0.9 (0.3)

3. Primary Outcome: Number of All Adverse Events Among the Participants With Mild Cognitive Impairment (MCI) Treated With Atomoxetine Compared to the Participants Treated With Placebo/Inactive Compound
Description: Safety was assessed by number of all adverse events among the participants treated with Atomoxetine compared to the participants treated with Placebo throughout the study. The Adverse Event assessment was done at each study visit through their participation in the study.
Time Frame: Up to Week 58
Population: In Atomoxetine/Placebo group 20 participants got Atomoxetine during period 1 and 18 got Placebo during period 2.
  In Placebo/ Atomoxetine group 19 participants got Placebo during period 1 and 19 participants got Atomoxetine during period 2.
  Total for Atomoxetine (20 in period 1 + 19 in period 2) Total for Placebo (19 in period 1+ 18 in period 2)
Measure: Number; unit: Adverse events
Groups:
- Atomoxetine: Participants in this arm received Atomoxetine, starting with 10 mg po daily and increasing weekly by increments to a maximum of 100 mg po daily or the maximum tolerated dose
- Inactive Compound (Placebo): Participants in this arm will receive a matching placebo that have inactive compound.
Arm/Group | Atomoxetine | Inactive Compound (Placebo)
Number analyzed (Participants) | 39 | 37
Adverse events | 142 | 91

4. Primary Outcome: Number of Participants That Drop Out of the Study Among the Participants Treated With Atomoxetine When Compared to the Participants Treated With Inactive Compound (Placebo)
Description: Tolerability is measured by comparing the drop out rate among the participants treated with Atomoxetine to the participants treated with inactive compound (Placebo). Study predicts that treatment-associated (Atomoxetine Group) drop out rate will be < 15% .
Time Frame: Up to Week 58
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Atomoxetine: Participants in this group received Atomoxetine starting with 10 mg po daily and increasing weekly by increments to a maximum of 100 mg po daily or the maximum tolerated dose.
- Inactive Compound/Placebo: Participants in this group received Matching placebo that have inactive compound.
Arm/Group | Atomoxetine | Inactive Compound/Placebo
Number analyzed (Participants) | 39 | 37
Participants | 2 | 1

5. Secondary Outcome: Rate of Cerebral Blood Flow in Subjects With Mild Cognitive Impairment MCI Treated With Atomoxetine / Inactive Compound Compared to Participants Treated With Inactive Compound / Atomoxetine
Description: Change in rate of cerebral blood flow is assessed by arterial spin labeling Magnetic Resonance Imaging (ASL-MRI) in subjects with Mild Cognitive Impairment MCI treated with Atomoxetine / Inactive Compound compared to participants treated with Inactive compound / Atomoxetine. The rates from the Baseline are compared to week 29 and week 58 among the participants treated with Atomoxetine / Inactive Compound compared to participants treated with Inactive compound / Atomoxetine. All MRIs will be reviewed by the investigators and the investigator.
Time Frame: Baseline, Week 29, Week 58
Population: This analysis includes participants who completed the entire study.
Measure: Mean (Standard Deviation); unit: mL/100 g/min
Arm/Group | Atomoxetine / Inactive Compound | Inactive Compound / Atomoxetine
Number analyzed (Participants) | 17 | 19
mL/100 g/min
  Baseline | 42.4 (8.6) | 42.6 (7.5)
  Week 29 | 39.3 (5.6) | 38.8 (6.2)
  Week 58 | 40.2 (7.1) | 39.6 (8.0)

6. Secondary Outcome: Change in FluoroDeoxyGlucose (FDG) Uptake in Participants With Mild Cognitive Impairment (MCI) Treated With Atomoxetine / Inactive Compound Compared to Participants Treated With Inactive Compound / Atomoxetine
Description: Cerebral metabolic rate for glucose as measured by Fluoro Deoxy Glucose (FDG) uptake will be obtained by Positron Emission Tomography (PET) scan. The rates from the Baseline are compared to week 29 and week 58 among the subjects treated with Atomoxetine / Inactive Compound Compared to Participants Treated With Inactive Compound / Atomoxetine. . Cerebral glucose metabolism is reduced in early stages of AD. The ratio of hippocampal FDG-PET uptake to the whole brain average are presented below.
Time Frame: Baseline, Week 29 and Week 58
Population: This analyses includes participants that completed 58 weeks of follow up.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Atomoxetine / Inactive Compound | Inactive Compound / Atomoxetine
Number analyzed (Participants) | 17 | 19
ratio
  Baseline | 0.69 (0.07) | 0.68 (0.08)
  Week 29 | 0.72 (0.08) | 0.67 (0.10)
  Week 58 | 0.74 (0.09) | 0.73 (0.08)

ADVERSE EVENTS:
Time Frame: All Adverse events were collected from Baseline to week 58 among the participants in both groups.
Groups:
- Atomoxetine: Participants in this arm included all the participants that received Atomoxetine, starting with 10 mg po daily and increasing weekly by increments to a maximum of 100 mg po daily or the maximum tolerated dose. The group includes 20 participants on Atomoxetine during period 1 and 19 participants on Atomoxetine during period 2.
- Inactive Compound: Participants in this arm included all the participants from both groups that received a matching placebo that have inactive compound. 19 participants on inactive compound during period 1 and 18 participants on inactive compound during period 2.
Arm/Group | Atomoxetine | Inactive Compound
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/37
Serious Adverse Events (participants affected / at risk) | 5/39 | 1/37
Other Adverse Events (participants affected / at risk) | 39/39 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=39) | Inactive Compound (N=37)
Fracture of Right Leg/Hip (Pelvis) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysautonomia (Nervous system disorders) | 1 (1) | 0 (0)
Hypothermia/dizziness (General disorders) | 1 (1) | 0 (0)
Headache Pain (General disorders) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Severe Elevated Blood Pressure (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=39) | Inactive Compound (N=37)
Headache (Vascular disorders) | 5 (7) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Falls (General disorders) | 6 (7) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (8)
Dizziness (General disorders) | 9 (11) | 8 (8)
Back Pain (General disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 2 (3) | 1 (2)
Loss of Appetite (General disorders) | 3 (3) | 0 (0)
Dry Mouth (General disorders) | 10 (10) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Suicide (General disorders) | 2 (2) | 1 (1)
Irritable Stomach (Gastrointestinal disorders) | 11 (14) | 5 (5)
Injury to Head and Ear (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 3 (3) | 3 (3)
Tremor (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Body Cramps (General disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Sample size is small leading to some analytical limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT01522404/Prot_SAP_000.pdf